CLINICAL TRIAL: NCT06900413
Title: Comparison of the Efficacy of Erector Spinae Plane (ESP) and External Oblique and Rectus Abdominis Plane (EXORA) Blocks in Laparoscopic Cholecystectomy
Brief Title: ESP vs. EXORA Blocks for Analgesia in Laparoscopic Cholecystectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aycan KURTARANGİL DOĞAN (Other)
Collaborators: Kutahya City Hospital (Other)
Responsible Party: Sponsor-Investigator, Aycan KURTARANGİL DOĞAN, Principal Investigator, Kutahya City Hospital
Organization: Kutahya City Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KSH-01
Record Dates: First submitted 2025-03-20; First posted 2025-03-28 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Erector Spinae Plane Block; Laparoscopic Cholecystectomy; Plane Block
Keywords: Erector Spinae Plane Block; exora block; laparoscopic cholecystectomy; patient-controlled analgesia; plane block

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group ESP (Active Comparator): The ESP block will be performed approximately 30 minutes before general anesthesia induction following sedation and standard monitoring. All block procedures will be conducted under sterile conditions, with skin preparation using dermol (%70 Isopropyl Alcohol, %2 Chlorhexidine Gluconate) and the ultrasound probe covered with a sterile drape.
  Interventions: Procedure: Group ESP
- Group EXORA (Active Comparator): The EXORA block will be performed 30 minutes before general anesthesia induction, following sedation and standard monitoring.
  Interventions: Procedure: Group EXORA

INTERVENTIONS:
Procedure: Group ESP — Experienced anesthesiologists with at least five years of expertise in regional anesthesia will perform the blocks under ultrasound guidance. A 4.0-12.0 MHz linear ultrasound probe (Affiniti 50; Philips) will be used. The ESP block will be applied at the T8 level on the right side, using an in-plane approach, while the patient is in a sitting position. The probe will be placed 2-3 cm lateral to the vertebra in a sagittal position to visualize the erector spinae muscle and transverse processes.
  A 22G, 100 mm block needle (Stimuplex® Ultra, Braun, Germany) will be advanced in a craniocaudal direction. The correct needle position will be confirmed by injecting 0.5-1 mL of isotonic NaCl and observing the spread via hydrodissection. Finally, 0.3 mL/kg of 0.25% bupivacaine will be administered, ensuring cranial and caudal spread of the local anesthetic.
  Arms: Group ESP
Procedure: Group EXORA — Experienced anesthesiologists with at least five years of expertise in regional anesthesia will administer the blocks under ultrasound guidance. A 4.0-12.0 MHz linear ultrasound probe will be placed laterally to the xiphoid process on the parasternal line in a sagittal position. The probe will be moved craniocaudally to identify the 6th rib and further advanced caudally to locate the 8th rib. Once the rectus abdominis muscle and 8th costal cartilage are identified, a 22G, 100 mm block needle will be used to administer 0.3 mL/kg of 0.25% bupivacaine. The correct spread of the local anesthetic will be confirmed via ultrasound.
  Arms: Group EXORA

SUMMARY:
Patients undergoing laparoscopic cholecystectomy may experience moderate to severe postoperative pain. Effective postoperative analgesia enhances patient comfort and accelerates recovery. This study aims to compare the effects of Erector Spinae Plane (ESP) and External Oblique and Rectus Abdominis Plane (EXORA) blocks on postoperative pain management and analgesic consumption.

The study is designed as a prospective, randomized, double-blind trial. Patients will be randomly assigned to groups, and both practitioners and evaluators will be blinded to group assignments. Our hypothesis is that the EXORA block will provide superior analgesia and require less analgesic consumption compared to the ESP block. The results will be assessed in terms of postoperative pain management, patient comfort, and additional analgesic requirements.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 65 years

Undergoing elective laparoscopic cholecystectomy

Classified as American Society of Anesthesiologists (ASA) physical status I to III

Providing written informed consent

Exclusion Criteria:

Known allergy or hypersensitivity to local anesthetics

Infection or skin lesions at the site of block application

Emergency surgical procedures

Refusal to participate in the study

Uncontrolled arterial hypertension

Uncontrolled diabetes mellitus

Mental retardation

Current use of antidepressant medications

Presence of metabolic disorders

Known bleeding diathesis

Morbid obesity (Body Mass Index > 40 kg/m²)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Tramadol consumption | 12 and 24 hours
  Total tramadol used in the first 12 and 24 hours postoperatively.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) for Pain Assessment | 30 minutes, 2 hours, 6 hours, 12 hours, and 24 hours after surgery
  Postoperative pain will be assessed using the Visual Analog Scale (VAS), which ranges from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate a worse outcome (more pain). Units on a scale (0-10)
Pinprick Sensory Block Test Results | 10 minutes, 20 minutes, and 30 minutes after the block, and 30 minutes after surgery
  Sensory block efficacy will be evaluated using the pinprick test at specified time intervals. The presence or absence of sensory block will be recorded. Binary (Block present / Block absent)
Nausea and Vomiting Score (NVS) | Within 24 hours after surgery
  Postoperative nausea and vomiting will be evaluated using the Nausea and Vomiting Scale (NVS), which includes:
  1. = No nausea,
  2. = Mild nausea,
  3. = Severe nausea,
  4. = Vomiting present. Higher scores indicate a worse outcome. Units on a scale (1-4)
Ramsay Sedation Scale (RSS) | Within 24 hours after surgery
  Postoperative sedation will be assessed using the Ramsay Sedation Scale (RSS), which includes:
  1. = Anxious, agitated, or restless
  2. = Cooperative, oriented, and tranquil
  3. = Responds to commands only
  4. = Brisk response to auditory stimulus
  5. = Sluggish response to auditory stimulus
  6. = No response Higher scores indicate a deeper level of sedation. Units on a scale (1-6)
Additional Analgesic Consumption | Within 24 hours after surgery
  The total amount of additional analgesics administered postoperatively will be recorded. Milligrams (mg)

OTHER OUTCOMES:
Total Antiemetic Consumption | Within 24 hours after surgery
  The total amount of antiemetic medication administered within 24 hours postoperatively will be recorded. Milligrams (mg)

CONTACTS AND LOCATIONS:
Overall Officials: Aycan KURTARANGİL DOĞAN, Principal Investigator — Kütahya City Hospital; Ali Kaynak, Principal Investigator — Kütahya City Hospital

IPD SHARING:
Plan to Share IPD: No